CLINICAL TRIAL: NCT00463294
Title: CABG Off or On Pump Revascularization Study (CORONARY)
Brief Title: Coronary Artery Bypass Surgery (CABG) Off or On Pump Revascularization Study
Acronym: CORONARY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: McMaster University (Other); University of Oxford (Other); Instituto Dante Pazzanese de Cardiologia (Other); Fu Wai Hospital, Beijing, China (Other); Universidad de La Frontera (Other); Fundación Cardiovascular de Colombia (Other); Charles University, Czech Republic (Other); Hopital Jean Minjoz (Other); Centre for Chronic Disease Control, India (Other); Ospedale Santa Croce-Carle Cuneo (Other); Medical University of Gdansk (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Ankara University (Other); Hotel Dieu Hospital (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other); SAL Hospital, Ahmedabad, India (Unknown)
Responsible Party: Principal Investigator, Andre Lamy, Cardiac Surgeon, Population Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRI-065
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: the Efficacy and Safety of Off-pump CABG
Keywords: CABG; On-pump; Off-pump
MeSH Terms: interventions — Coronary Artery Bypass; Coronary Artery Bypass, Off-Pump

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- On Pump Arm (Active Comparator)
  Interventions: Procedure: Coronary Artery Bypass Graft with the use of CPB
- Off Pump Arm (Experimental)
  Interventions: Procedure: Coronary Artery Bypass Graft without the use of CPB

INTERVENTIONS:
Procedure: Coronary Artery Bypass Graft with the use of CPB — Coronary Artery Bypass Graft (CABG) using median sternotomy, CPB, cardioplegia and complete cross-clamp and no associated or concomitant surgical procedures
  Other Names: ON Pump CABG
  Arms: On Pump Arm
Procedure: Coronary Artery Bypass Graft without the use of CPB — Coronary Artery Bypass Graft (CABG) with no associated or concomitant surgical procedures, using median sternotomy and without CPB and cardioplegia
  Other Names: OFF Pump
  Arms: Off Pump Arm

SUMMARY:
I. Main Research Question:

* To compare the risks and benefits of Off-pump Coronary artery bypass surgery (CABG) to On-pump CABG and to determine if one is better than the other.
* The purpose of this pilot study is also to see the rate of recruitment with expertise-based randomization across different hospital settings.

II. Small RCT studies and meta-analyses done so far have not been able to conclusively say which of the procedure is better. A large randomized study is required to establish the risks and benefits associated with both the off-pump and on-pump CABG surgical procedures.

III. The study will look at which of the two techniques reduce major risks associated with CABG.

DETAILED DESCRIPTION:
Rationale and purpose of the study:

Coronary artery bypass grafting (CABG) surgery prolongs life-expectancy in patients with severe ischemic heart disease, especially those with left main, triple vessel disease or single/double vessel disease with stenosis of the proximal left anterior descending (LAD) artery. The perioperative mortality is about 2% with an additional 5% to 7% suffering complications such as myocardial infarction, stroke, renal failure, etc. The technique of operating on a beating heart (off-pump) for coronary artery bypass grafting surgery has been recently developed in the past few years in an effort to decrease the above perioperative complications typically related to cardiopulmonary bypass associated with on-pump CABG. While registries suggest that off-pump CABG may be superior, these data cannot fully control for differences in patient characteristics, which influence patient selection for specific procedures. The benefits of off-pump CABG compared with conventional on-pump CABG are unclear. The investigators therefore propose a large simple, international multicentre randomized controlled trial to definitively evaluate the efficacy and safety of off-pump CABG in the treatment of patients undergoing coronary artery surgery funded by CIHR, this pilot study will be a preliminary step towards a full trial.

Sample size:

The investigators examined the outcomes in the Canadian off-pump CABG Registry to identify a group of patients who represent a higher risk of cardiovascular events. Utilizing the inclusion criteria described below, this group of patients has accumulated the vast majority of outcomes in the Registry and represent more than 50% of patients in the Registry, therefore minimizing the sample size but still being representative. The cumulative event rate at 30 days (first co-primary outcome) for on-pump CABG is estimated as being 8.6% and the investigators expect a 33% relative risk reduction (RRR) for the off-pump CABG group. The sample calculated for the whole trial is 4700 patients.

Design/Methodology:

Trial design: This is a pilot randomized controlled trial comparing off-pump CABG versus on-pump CABG in 60 patients who will be undergoing isolated CABG.

Interventions: Patients eligible for CABG will be randomized to receive either an Off-pump CABG surgery or On-pump CABG surgery.

Randomization: After obtaining informed written consent patients will be allocated to either off-pump CABG or on-pump CABG by calling a 24-hour randomization telephone number. An expertise-based randomization will be used wherein a surgeon who is an expert in Off-pump surgery will operate on patients randomized to receive Off-pump surgery. Patients randomized to receive On-pump CABG will be operated on by a surgeon who is an expert in on-pump CABG surgery. To minimize bias stratified block randomization will used. For this pilot study randomization will be stratified to 3 centres and random block of 4 or 6.

The data adjudicators will be blinded to the study. Due to the nature of intervention, the operating surgeon, anesthetist, perfusionist, other operation room staff, intensive-care unit staff will not be blinded in this study.

Setting:

Patients will have either been seen in the emergency, outpatient or ICU and diagnosed with having single, double or triple coronary artery occlusion requiring an isolated CABG.

Study interventions:

Interventions: Patients eligible for CABG will be randomized to receive either an Off-pump CABG surgery or On-pump CABG surgery. A surgeon who is an expert in the assigned technique will perform the procedure.

Primary outcomes:

* The occurrence of the composite of total mortality, stroke, nonfatal MI, or new renal failure at 30 days post CABG surgery AND
* The occurrence of the composite of total mortality, stroke, nonfatal MI, new renal failure, or repeat coronary revascularization (i.e. coronary artery bypass surgery or percutaneous coronary intervention) over 5 years after randomization.

The secondary outcomes

* The assessment of total costs and resources consumption at 30 days after CABG surgery AND
* The assessment of total costs and resources consumption at 5 years after CABG surgery

Measurements:

The investigators will ascertain all events of interest through periodic and regular follow-up utilizing standardized definitions for all events, appropriate supporting documents will be obtained centrally.

* CV death: all deaths are considered cardiovascular unless a specific non-cardiovascular cause is evident (e.g. malignancy).
* Stroke: new acute focal neurological deficit (except for subarachnoid hemorrhage which may not be focal) thought to be of vascular origin with signs or symptoms lasting greater than 24 hours.
* MI perioperative (within 24 hours of surgery): new pathologic Q waves with documented new wall motion abnormalities other than septal OR cardiac markers ³ 10 x ULN.
* MI non-perioperative (later than 24 hours after surgery): ECG changes consistent with infarction (new significant Q waves in two contiguous leads in the absence of previous LVH or conduction abnormalities) or evolving ST-segment to T-wave changes in two contiguous leads or new left bundle branch block or ST segment elevation requiring thrombolysis or PCI AND cardiac markers (troponins or CKMB) in the necrosis range. Post-PCI MI are included into non-perioperative MI group but are defined as new pathologic Q waves with documented new wall motion abnormalities other than septal OR cardiac markers ³ 3 x ULN within 24 hours of PCI.
* Renal failure: doubling of serum creatinine from pre-op baseline or requirement for renal replacement therapy (eg, dialysis, continuous hemofiltration, renal transplant). Hemofiltration or dialysis only during cardio-pulmonary bypass does not constitute a requirement for renal replacement therapy. Patients who receive dialysis within 1 month of the surgery are not eligible for this endpoint.
* Repeated coronary revascularization: new CABG procedure or PCI associated with documented ischemia by stress testing (ECG, ECHO, or nuclear) AND graft failure or new culprit lesion (³ 70% luminal stenosis).

For other endpoints, the investigators have defined:

* Recurrence of angina: new or chronic onset of typical chest pain with documented ischemia by stress testing (ECG, ECHO, or nuclear).
* Blood transfusions: all blood bank products transfused within 24 hours of the CABG surgery.
* Total mortality: all causes of mortality

Plan for data analysis:

The intention to treat principle, in which all participants will be included in their assigned treatment groups regardless of adherence, will guide all analyses. In the principle analysis, the time to the first occurrence of one of the components of the cluster of (cardiac death, stroke, nonfatal MI, new renal failure) will be presented by Kaplan-Meier survival curves and the comparisons between the two treatment groups will be performed by a log-rank test. The treatment effect as measured by the hazard ratio and 95% confidence interval will be derived by the Cox proportional hazards model. The investigators will also calculate the absolute risk reductions and the associated 95% confidence intervals, as well as the number needed to treat (NNT) with off-pump CABG to prevent one major cardiovascular event. Participants who prematurely discontinue follow-up before a major cardiovascular event will be censored as to their last follow-up data; this number is expected to be <1% given the relatively short period of follow-up after surgery.

In secondary analyses the investigators will determine and compare the incidence of major cardiovascular events (cardiac death, stroke, nonfatal MI, new renal dialysis) and revascularization procedures (i.e. coronary artery bypass surgery and percutaneous coronary intervention) using the same strategy. The effect of the two operative techniques on different sub-groups (i.e. patients with diabetes, renal failure, congestive heart failure, cerebrovascular disease, as well as patient left ventricular function, gender and ages will be conducted by stratified analysis through a Cox proportional hazards model. The test of interaction between each subgroup factor and the treatment group will be done by including a product term in the model already containing treatment and the subgroup factor. The length of hospital stay and length of ICU/CCU stay will be compared using a student's t-test. An events adjudication committee (blind to surgical allocation) will centrally review all suspected major outcomes listed above.

The investigators will also do subgroup analysis on different sub-groups (i.e. patients with diabetes, renal failure, congestive heart failure, cerebrovascular disease, as well as patient left ventricular function, gender and ages will be examined for consistency and coherence)

ELIGIBILITY:
Inclusion Criteria:

Patients who have been diagnosed with coronary artery disease (single, double or triple disease) will be eligible if they:

1. require isolated CABG with median sternotomy
2. are able to give their informed written consent
3. are> 21 years of age and
4. have one or more of the following risk factors:

   * ≥ 70 years
   * peripheral vascular disease (previous peripheral bypass or amputation or ABI <0.80)
   * Cerebrovascular disease (history of stroke, TIA)
   * Renal insufficiency (creatinine above upper limit of normal)
   * >60 years of age and one of the following:

     * diabetes (oral hypoglycemic agent and/or insulin)
     * urgent revascularization (waiting in hospital)
     * LV ejection fraction <35%
     * current or recent smoker.
   * 55-59 years of age and two of the following:

     * diabetes (oral hypoglycemic agent and/or insulin)
     * urgent revascularization (waiting in hospital)
     * LV ejection fraction <35%
     * current or recent smoker.

Exclusion Criteria:

Patients will be excluded if they have one of the following:

1. concomitant cardiac procedure associated with CABG,
2. contra-indications to off-pump CABG or on-pump CABG (calcified aorta, intramuscular LAD, calcified coronaries, small target vessels)
3. concomitant life-threatening disease likely to limit life expectancy to less than 2 years,
4. prior enrollment in this trial
5. emergency CABG surgery (immediate revascularization for hemodynamic instability) OR
6. redo CABG.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4752 (Actual)
Dates: Start 2007-10; Primary Completion 2012-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
First Co-Primary Outcome | 30 days post CABG surgery
  The occurrence of the composite of total mortality, stroke, nonfatal MI, or new renal failure at 30 days post CABG surgery
Second co-primary outcome | 5 years after CABG
  The occurrence of the composite of total mortality, stroke, nonfatal MI, new renal failure, or repeat coronary revascularization (i.e. coronary artery bypass surgery or percutaneous coronary intervention) over 5 years after randomization.

SECONDARY OUTCOMES:
The assessment of total costs and resources consumption at 30 days after CABG surgery | 30 days after CABG surgery
The assessment of total costs and resources consumption at 5 years after CABG surgery | 5 years after CABG surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lamy Andre, MD, MSc, Principal Investigator — McMaster University; Salim Yusuf, MD, DPhil, Principal Investigator — Population Health Research Institute; David Taggart, MD, Principal Investigator — University of Oxford
Locations (52):
- Fundacion Medica de rio negro y neuquen, Rio Negro, Argentina
- Brazil (11):
  - Beneficencia Portuguesa de Sao Paulo, São Paulo, CEP
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, CEP
  - Hospital Sao Francisco Complexo Hospitalar Santa Casa, Porto Alegre, Rio Grande do Sul
  - Irmande Santa Casa De Misericordia De Curtiba, Curitiba Parana
  - Braile Clinica de Servicos de Assistencia Medico, São José do Rio Preto
  - Irmandade da Santa Casa de Misericordia de Sao Paulo, São Paulo
  - Federal University of Sao Paulo School of Medicine, São Paulo
  - Associação do Sanátorio Sírio, São Paulo
  - Instituto do Coracao do Hospital das Clinicas da, São Paulo
  - Hospital Mario Covas, São Paulo
  - Santa Casa de Misericordia de Marilia, São Paulo
- Canada (6):
  - Foothills Medical Centre, Calgary, Alberta
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Hotel-Dieu du CHUM, Montreal, Quebec
- Chile (2):
  - Hospital Regional Temuco, Temuco, Región de la Araucanía
  - Instituto Nacional del Torax, Santiago
- China (3):
  - ChaoYang Hospital, Beijing
  - FuWai Hospital, Beijing
  - Nanjing First Hospital, Nanjing
- Colombia (2):
  - Fundacion Cardioinfantil, Bogotá
  - Fundacion Valle Del Lili, Cali
- Czechia (6):
  - Charles University Hospital, Hradec Králové
  - Kardiochirurgicke centrum, Ostrava-Poruba
  - University Hospital Pilsen, Pilsen
  - Fakultni nemocnice Kralovske Vinohrady (FNKV), Prague
  - University Hospital Motol, Prague
  - Nemocnice Podlesi, Třinec
- Service de chirurgie thoracique et cardio-vasculaire, Besançon, France
- India (9):
  - Nizam's Institute of Medical Sciences, Hyderabad, Andhra Pradesh
  - SAL Hospital and Medical Institute, Ahmedabad, Gujarat
  - Amrita Institute of Medical Sciences and Research Center, Kochi, Kerala
  - G.Kuppuswamy Naidu Memorial Hospital, Coimbatore, Tamil Nadu
  - SAL Hospital, Ahmedabad
  - International Center of Cardiovascular and Thoracic Diseases, Chennai Tamil Nadu
  - Sanjay Gandhi PGIMS, Lucknow
  - All India Institute of Medical Sciences, New Delhi
  - Escorts Heart Institute and Research Centre, Noida
- Italy (2):
  - Ospedale S. Croce, Cuneo
  - Ospedale Niguarda - Ca Granda, Milan
- Jagiellonian University, Krakow, Poland
- Turkey (Türkiye) (5):
  - Alp Aslan, Ankara
  - Erol Senor, Ankara
  - Ruchan Akar, Ankara
  - Sertap Aykut Aka, Ankara
  - Volkan Sinci, Ankara
- United Kingdom (3):
  - Basildon and Thurrock University Hospital NHS FT, Basildon, Essex
  - Royal Infirmary of Edinburgh, Edinburgh, EU
  - The John Radcliffe Hospital, Oxford

REFERENCES:
- [Derived] Dimagli A, Gaudino M, An KR, Olaria RP, Soletti GJ, Cancelli G, Harik L, Noiseux N, Stevens LM, Lamy A; CORONARY investigators. Five-Year Hospital Readmission After Coronary Artery Bypass Surgery and the Association With Off-Pump Surgery and Sex. J Am Heart Assoc. 2023 Apr 18;12(8):e028063. doi: 10.1161/JAHA.122.028063. Epub 2023 Apr 7. PMID 37026546
- [Derived] Hebert M, Lamy A, Noiseux N, Stevens LM; CORONARY Investigators. Impact of early quantitative morbidity on 1-year outcomes in coronary artery bypass graft surgery. Interact Cardiovasc Thorac Surg. 2022 Mar 31;34(4):523-531. doi: 10.1093/icvts/ivab316. PMID 34788466
- [Derived] Conen D, Wang MK, Devereaux PJ, Whitlock R, McIntyre WF, Healey JS, Yuan F, Yusuf S, Lamy A. New-Onset Perioperative Atrial Fibrillation After Coronary Artery Bypass Grafting and Long-Term Risk of Adverse Events: An Analysis From the CORONARY Trial. J Am Heart Assoc. 2021 Jun 15;10(12):e020426. doi: 10.1161/JAHA.120.020426. Epub 2021 May 29. PMID 34056913
- [Derived] Lamy A, Devereaux PJ, Prabhakaran D, Taggart DP, Hu S, Straka Z, Piegas LS, Avezum A, Akar AR, Lanas Zanetti F, Jain AR, Noiseux N, Padmanabhan C, Bahamondes JC, Novick RJ, Tao L, Olavegogeascoechea PA, Airan B, Sulling TA, Whitlock RP, Ou Y, Gao P, Pettit S, Yusuf S; CORONARY Investigators. Five-Year Outcomes after Off-Pump or On-Pump Coronary-Artery Bypass Grafting. N Engl J Med. 2016 Dec 15;375(24):2359-2368. doi: 10.1056/NEJMoa1601564. Epub 2016 Oct 23. PMID 27771985
- [Derived] Lamy A, Tong W, Devereaux PJ, Gao P, Gafni A, Singh K, Taggart D, Straka Z, Akar AR, Piegas L, Ou Y, Yusuf S. The cost implications of off-pump versus on-pump coronary artery bypass graft surgery at one year. Ann Thorac Surg. 2014 Nov;98(5):1620-5. doi: 10.1016/j.athoracsur.2014.06.046. Epub 2014 Sep 24. PMID 25261272
- [Derived] Garg AX, Devereaux PJ, Yusuf S, Cuerden MS, Parikh CR, Coca SG, Walsh M, Novick R, Cook RJ, Jain AR, Pan X, Noiseux N, Vik K, Stolf NA, Ritchie A, Favaloro RR, Parvathaneni S, Whitlock RP, Ou Y, Lawrence M, Lamy A; CORONARY Investigators. Kidney function after off-pump or on-pump coronary artery bypass graft surgery: a randomized clinical trial. JAMA. 2014 Jun 4;311(21):2191-8. doi: 10.1001/jama.2014.4952. PMID 24886787
- [Derived] Lamy A, Devereaux PJ, Prabhakaran D, Taggart DP, Hu S, Paolasso E, Straka Z, Piegas LS, Akar AR, Jain AR, Noiseux N, Padmanabhan C, Bahamondes JC, Novick RJ, Vaijyanath P, Reddy SK, Tao L, Olavegogeascoechea PA, Airan B, Sulling TA, Whitlock RP, Ou Y, Pogue J, Chrolavicius S, Yusuf S; CORONARY Investigators. Effects of off-pump and on-pump coronary-artery bypass grafting at 1 year. N Engl J Med. 2013 Mar 28;368(13):1179-88. doi: 10.1056/NEJMoa1301228. Epub 2013 Mar 11. PMID 23477676
- [Derived] Garg AX, Devereaux PJ, Yusuf S, Cuerden MS, Parikh CR, Coca SG, Walsh M, Cook RJ, Whitlock RP, Noiseux N, Novick RJ, Ou Y, Lamy A; CORONARY Investigators. Coronary Artery Bypass Grafting Surgery Off- or On-pump Revascularisation Study (CORONARY): kidney substudy analytic protocol of an international randomised controlled trial. BMJ Open. 2012 Apr 18;2(2):e001080. doi: 10.1136/bmjopen-2012-001080. Print 2012. PMID 22514244
- [Derived] Lamy A, Devereaux PJ, Prabhakaran D, Taggart DP, Hu S, Paolasso E, Straka Z, Piegas LS, Akar AR, Jain AR, Noiseux N, Padmanabhan C, Bahamondes JC, Novick RJ, Vaijyanath P, Reddy S, Tao L, Olavegogeascoechea PA, Airan B, Sulling TA, Whitlock RP, Ou Y, Ng J, Chrolavicius S, Yusuf S; CORONARY Investigators. Off-pump or on-pump coronary-artery bypass grafting at 30 days. N Engl J Med. 2012 Apr 19;366(16):1489-97. doi: 10.1056/NEJMoa1200388. Epub 2012 Mar 26. PMID 22449296
- [Derived] Lamy A, Devereaux PJ, Prabhakaran D, Hu S, Piegas LS, Straka Z, Paolasso E, Taggart D, Lanas F, Akar AR, Jain A, Noiseux N, Ou Y, Chrolavicius S, Ng J, Yusuf S. Rationale and design of the coronary artery bypass grafting surgery off or on pump revascularization study: a large international randomized trial in cardiac surgery. Am Heart J. 2012 Jan;163(1):1-6. doi: 10.1016/j.ahj.2011.10.007. PMID 22172429